CLINICAL TRIAL: NCT06393621
Title: Prospective, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Proof-of-Concept Study to Investigate the Effectiveness of KEFPEP® on Regulating High Blood Pressure
Brief Title: Investigate the Effectiveness of KEFPEP® on Regulating High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Chung Hsing University (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Chuan -Mu Chen, Chair Professor, National Chung Hsing University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHP1705H01; 201707074MIPC (Other: NTUH-REC)
Record Dates: First submitted 2024-03-20; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Prehypertension
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KEFPEP® (Experimental): 1. Dosage form: Powder (directly take the powder with appropriate amount of warm water)
  2. Dose(s): Total 2.8 g kefir-fermented milk powder with increased peptide content 1.2 g.
  Interventions: Dietary Supplement: KEFPEP®
- Placebo (Placebo Comparator): 1. Dosage form: Powder (directly take the powder with appropriate amount of warm water).
  2. Dose(s): Total 2.8 g starch power.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: KEFPEP® — Twice daily (one pack before breakfast and the other before dinner)
  Arms: KEFPEP®
Other: Placebo — Twice daily (one pack before breakfast and the other before dinner)
  Arms: Placebo

SUMMARY:
To assess the ability of KEFPEP® to reduce blood pressure

DETAILED DESCRIPTION:
Primary objective-

• To assess the ability of KEFPEP® to reduce blood pressure.

Secondary objective-

1. To access the effect of KEFPEP® on vascular inflammation or damage.
2. To access the effect of KEFPEP® on cardiovascular diseases prevention.
3. To assess the safety of KEFPEP® .

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ages 20 years or older.
2. Belong to either one of the following categories based on the Seventh Report of the Joint National Committee (JNC 7) as measured by office BP at Screening visit:

   * Prehypertension (SBP 120 - 139 mmHg or DBP 80 - 89 mmHg)
   * Stage I hypertension (SBP 140 - 159 mmHg or DBP 90 - 99 mmHg)
3. Body weight≤90 kg, and BMI≥18.5 kg/m2 or < 30 kg/m2.
4. NOT on any antihypertensive treatment at the time of entry into the study.
5. Willing to comply with the study procedures and follow-ups.
6. Understand the nature of the study, and have signed informed consent forms.

Exclusion Criteria:

1. Patients with any of the following conditions within 6 months prior to study participation:

   * Secondary hypertension
   * Uncontrolled diabetes mellitus
   * Renal disease based on the investigator's judgment
   * Severe hepatic disease with Child-Pugh class C
   * Severe anaemia
   * Any malignant disease or serious disease
2. Patients with clinically significant abnormalities in the following laboratory parameters within 2 weeks prior to Screening visit or during the screening period:

   * HbA1c > 9%
   * AST or ALT ≥ 3 x upper limit of normal (ULN)
   * Estimated glomerular filtration rate (eGFR) < 50 ml/min/1.73 m2
   * Serum creatinine ≥ 3 x ULN
   * Hemoglobin < 10 g/dL
3. History of milk allergy and/or lactose intolerance.
4. History of alcohol abuse.
5. Constant use of oral medication or supplements affecting blood pressure.
6. Female patients who are pregnant, planning to become pregnant, or lactating.
7. Male or female patients of child-bearing potential do not agree to use an effective method of contraception during the study period.
8. Currently participating in any other interventional clinical study within 30 days
9. Patients who are considered not suitable for the study according to the investigator's judgment for the patient's best interest.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Reduction of 5 mmHg SBP | At week 12
  I. Reduction of 5 mmHg from Baseline in office SBP. II. Reduction of 5 mmHg from Baseline in 24-hour ambulatory SBP.
Reduction of 10 mmHg SBP | At week 12
  I. Reduction of 10 mmHg from Baseline in office SBP. II. Reduction of 10 mmHg from Baseline in 24-hour ambulatory SBP.

SECONDARY OUTCOMES:
Office SBP and diastolic blood pressure (DBP) | Baseline (Day 1/Visit 3), Week 4 (Visit 4), Week 8 (Visit 5), and Week 12 (Visit 6)
  Compare the change from Baseline in office SBP and DBP
24-hour ambulatory | Baseline (Day 1/Visit 3) and Week 12 (Visit 6)
  Compare the change from Baseline in 24-hour ambulatory SBP and 24-hour ambulatory DBP
Biomarkers of blood vessel inflammation | Baseline (Day 1/Visit 3) and Week 12 (Visit 6)
  Biomarker: high sensitivity C-Reactive Protein (hsCRP); Unit of Measure: mg/L (milligrams per liter). By separating these biomarkers into distinct outcome measures, it ensures clarity in reporting and analysis, especially when different units of measure are involved.
Biomarkers of blood vessel damage | Baseline (Day 1/Visit 3) and Week 12 (Visit 6)
  Biomarker: creatine kinase; Unit of Measure: U/L (unit per liter). By separating these biomarkers into distinct outcome measures, it ensures clarity in reporting and analysis, especially when different units of measure are involved.
Follow-up and safety analyses -Vital signs | The 2-week follow-up period once completing the 12-week dietary
  Measure the subject's body temperature (°C), respiratory rate per minute, and heartbeat/pulse per minute.
  (Measured the subject's sitting office blood pressure at revisit. At each measurement, the subject should rest in an air-conditioned space for approximately 30 minutes until the blood pressure stabilizes before using an electronic sphygmomanometer to measure the blood pressure while seated. The subject's body temperature (°C), respiratory rate per minute, and heartbeat/pulse per minute were displayed simultaneously in the electronic blood pressure monitor.)
Follow-up and safety analyses -Adverse events (AEs) | The 2-week follow-up period once completing the 12-week dietary
  Adverse events were according to MedDRA version 26.0, and all events were classified according to Preferred Terms (PT) and System Organ Class (SOC).

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Kuang Lee, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Cholongitas E, Papatheodoridis GV, Vangeli M, Terreni N, Patch D, Burroughs AK. Systematic review: The model for end-stage liver disease--should it replace Child-Pugh's classification for assessing prognosis in cirrhosis? Aliment Pharmacol Ther. 2005 Dec;22(11-12):1079-89. doi: 10.1111/j.1365-2036.2005.02691.x. PMID 16305721
- [Background] Chronic kidney disease in adults: assessment and management. London: National Institute for Health and Care Excellence (NICE); 2015 Jan. Available from http://www.ncbi.nlm.nih.gov/books/NBK555204/ PMID 32208570

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT06393621/Prot_ICF_000.pdf